CLINICAL TRIAL: NCT05142202
Title: Doubly Accelerated Partial Breast Irradiation After Breast-Conserving Surgery for Early Breast Cancer - High Five (HiFi) APBI Study
Brief Title: High Five (HiFi) Accelerated Partial Breast Irradiation Study
Acronym: HiFi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Greater Poland Cancer Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HiFi-APBI
Record Dates: First submitted 2021-11-08; First posted 2021-12-02 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; breast-conserving surgery; brachytherapy; High Five; APBI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Doubly Accelerated Partial Breast Irradiation after Breast-Conserving Surgery (Experimental): All recruited participants will be treated with adjuvant to breast-conserving surgery accelerated partial breast irradiation with multicatheter interstitial brachytherapy technique and prescribed five times 5,4 Gy delivered in 3 consecutive days (6 hours minimum gap between the fractions). Treatment starts not later than 12 weeks after surgery (optimally 4-8 weeks), after wound healing, and obtaining the final pathological report with full immunohistochemistry and proper risk group assignment.
  The control group consists of standard adjuvant APBI with multicatheter interstitial brachytherapy technique 8 x 4 Gy in 5 consecutive days or 7 x 4,3 Gy in 4 consecutive days (6 hours minimum gap between the fractions).
  Interventions: Radiation: Breast Irradiation after Breast-Conserving Surgery

INTERVENTIONS:
Radiation: Breast Irradiation after Breast-Conserving Surgery — All recruited participants will be treated with adjuvant to breast-conserving surgery accelerated partial breast irradiation with multicatheter interstitial brachytherapy technique and prescribed five times 5,4 Gy delivered in 3 consecutive days (6 hours minimum gap between the fractions). Treatment starts not later than 12 weeks after surgery (optimally 4-8 weeks), after wound healing, and obtaining the final pathological report with full immunohistochemistry and proper risk group assignment.

SUMMARY:
To establish the role of adjuvant multicatheter interstitial high-dose-rate brachytherapy in doubly accelerated and radiobiologically equivalent irradiation scheme of 5 x 5,4 Gy in 3 days of treatment (High Five, HiFi-APBI) compared to the adopted long-term standard of APBI realized in 4-5 days (7-8 x 4-4,3 Gy) in selected women with breast low-risk invasive cancer or carcinoma in-situ, in terms of 3-month early and 2-year late toxicity.

DETAILED DESCRIPTION:
Early low-risk breast cancer treatment with high-dose-rate brachytherapy (HDR-BT) (according to GEC-ESTRO, ASTRO, ABS recommendations) as a sole adjuvant treatment to the tumor bed after breast-conserving surgery (BCS) is acknowledged by prominent oncological societies in Poland and the world (PTB - Polish Brachytherapy Society, PTRO - Polish Society for Radiation Oncology, PTO - Polish Society of Oncology, ESTRO, ABS, ASTRO, ASCO). Treatment with multicatheter interstitial HDR-BT in the form of accelerated partial breast irradiation (APBI) was successfully verified in multi-institutional randomized clinical trials (Hungarian trial, GEC-ESTRO trial). It defined the currently widely used oncologically effective and clinically safe irradiation scheme of 8 x Gy in 5 days or 7 x 4,3 Gy in 4 days. In the USA, the irradiation scheme of 10 x 3,4 Gy is widely used in 5-10 days (e.g., NSABP-B39). Some European and American centers are investigating and publishing preliminary results of extremely shortened irradiation schemes of 4 x 6,25 Gy or 3 x 7,5 Gy in 2-3 treatment days, perioperatively (vAPBI trial - Valencia, TRIUMPH-T trial - Phoenix). In the Brachytherapy Department at Greater Poland Cancer Center (GPCC), the listed regimen of 7-8 x 4-4,3 Gy in 4-5 days has been used successfully since 2008. It results in very high local control rates and very low radiation-induced toxicity. APBI after BSC ensures, in properly selected low-risk patients, an equivalent local control rate and lower toxicity compared to whole breast irradiation with external beam radiation therapy (EBRT) The study hypothesis is that an additional moderately shortened irradiation scheme of 5 x 5,4 Gy in 3 consecutive days (two fractions daily with minimal 6 hours gap between fractions) does not increase early toxicity and 2-years late toxicity (primary endpoint). Also, it ensures the same or potentially higher 2-years local control probability compared to the standard regimen (control group).

What is essential, all the above-listed regimens are equivalent in terms of EQD2 calculations. The advantage of higher fraction doses that enable scheme shortening is relatively low radiobiological α/β ratio, estimated for breast cancer at around 4.

The study's primary goal is to prove the possibility of further gradual shortening of the total time of postoperative adjuvant treatment, thus, in the face of increasing breast cancer morbidity, increasing its accessibility. Indirectly, the shortened regimen may decrease the financial burden of the patient and the health system, reduce the patient's oncological treatment-related stress, absence from work, and separation from family. The project feasibility is likely since the only difference between standard and experimental procedures is in the dose and its number.

It's a prospective mono-institutional non-randomized open-label pilot study which results would be a base for further research on larger patients' groups in an anticipated multi-institutional randomized study.

The primary endpoint is to establish the role of adjuvant HDR brachytherapy in the allowable doubly accelerated and radiobiologically equivalent irradiation scheme of 5 x 5,4 Gy in 3 days of treatment (High Five, HiFi-APBI) compared to the adopted long-term standard of APBI realized in 4-5 days (7-8 x 4-4,3 Gy) in patients with breast low-risk invasive cancer or carcinoma in-situ, in terms of 3-month early and 2-year late toxicity.

Secondary endpoints: 1. Assessment of 2-years local control rate; 2. Review of 2-years cosmetic result; 3. Evaluation of the quality of life (QOL); 4. Evaluation of the overall survival (OS), disease-free survival (DFS), and distant metastases free survival (DFMS); 5. Analysis of the performed surgical approaches (tumorectomy, quadrantectomy, oncoplasty) preceding HDR-BT and their influence on the cosmetic results.

It is assumed to recruit a minimum of 60 participants in 2-3 years. The historical control group from the last three years counts over a hundred patients. The study is planned to be continued for up to 5 years to reach a substantially extended follow-up of 2 years.

Assumed causes of study termination: the occurrence of two or more cases of the treated area fat necrosis in which surgical intervention would be necessary (conservative treatment ineffective); too low recruitment (less than one-third of planned); occurrence of two or more similar and earlier not observed cases.

ELIGIBILITY:
Inclusion Criteria:

* stage 0-II breast cancer
* Invasive ductal carcinoma (NOS, NST, other subtypes), invasive lobular carcinoma, ductal carcinoma in situ (DCIS)
* Invasive carcinoma/DCIS, which is unifocal and unicentric
* pT1-2, maximal tumor size < 3 cm
* pN0 (no metastases to the nodes)
* LVI(-) - no lymphovascular invasion
* M0 (no distant metastases)
* Surgical margins free of cancer (no tumor on ink) in each direction; in the case of DCIS, the minimum margin of 2 mm in each direction
* Lack of indications to chemotherapy/immunotherapy pre- or postsurgically (e.g., triple-negative, HER2-positive breast cancer)
* Treatment start not later than 12 weeks after surgery (optimally 4-8 weeks, after wound healing)
* Informed handwritten signed patient's consent

Exclusion Criteria:

* stage III-IV breast cancer
* pT2-4, maximal tumor size ≥ 3 cm
* surgical margins cannot be properly microscopically assessed
* EIC(+) - presence of extensive intraductal component
* Paget's disease or microscopically assessed skin involvement
* pN1-3M1 (presence of nodal or distant metastases)
* pre- or postsurgical indications for chemotherapy/immunotherapy
* other cancer (less than five years at time of recruitment) except skin cancer or cured FIGO 0-I cervical cancer
* time of pregnancy or lactation
* collagen disorders (congenital or acquired)
* psychiatric disorder disabling patient's compliance
* breast appearance or postsurgical status disabling safe interstitial multicatheter implantation
* lack of informed handwritten signed patient's consent

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 50 years, postmenopausal
Enrollment: 147 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adjuvant treatment - the early toxicity incidence | Up to 48 months
  The early toxicity incidence (radiodermatitis, hematoma, breast infection, intraoperative breast damage, breast pain) according to the Common Terminology Criteria for Adverse Events v5.0 (CTCAE) in 3 months frame.
Adjuvant treatment - the late toxicity incidence | up to 48 months
  The late toxicity incidence (skin, subcutaneous tissue) according to the RTOG/EORTC Late Radiation Morbidity Scoring Schema in 24 months frame.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Chicheł, PhD, MD, Principal Investigator — Greater Poland Cancer Centre
Locations (1):
- Greater Poland Cancer Centre, Poznan, Greater Poland Voivodeship, Poland

REFERENCES:
- [Background] Guinot JL, Gonzalez-Perez V, Meszaros N, Major T, Najjari-Jamal D, Gutierrez-Miguelez C, Santos MA, Smanyko V, Laplana M, Polgar C; GEC-ESTRO Breast Working Group2. Very accelerated partial breast irradiation Phase I-II multicenter trial (VAPBI): Feasibility and early results. Brachytherapy. 2021 Mar-Apr;20(2):332-338. doi: 10.1016/j.brachy.2020.10.010. Epub 2020 Nov 19. PMID 33223449
- [Background] Hannoun-Levi JM, Lam Cham Kee D, Gal J, Schiappa R, Hannoun A, Fouche Y, Gautier M, Boulahssass R, Chand ME. Accelerated partial breast irradiation in the elderly: 5-Year results of the single fraction elderly breast irradiation (SiFEBI) phase I/II trial. Brachytherapy. 2020 Jan-Feb;19(1):90-96. doi: 10.1016/j.brachy.2019.10.007. Epub 2019 Nov 23. PMID 31767533
- [Background] Khan AJ, Chen PY, Yashar C, Poppe MM, Li L, Abou Yehia Z, Vicini FA, Moore D, Dale R, Arthur D, Shah C, Haffty BG, Kuske R. Three-Fraction Accelerated Partial Breast Irradiation (APBI) Delivered With Brachytherapy Applicators Is Feasible and Safe: First Results From the TRIUMPH-T Trial. Int J Radiat Oncol Biol Phys. 2019 May 1;104(1):67-74. doi: 10.1016/j.ijrobp.2018.12.050. Epub 2019 Jan 4. PMID 30611839
- [Background] Rivera S, Hannoun-Levi JM. Hypofractionated radiation therapy for invasive breast cancer: From moderate to extreme protocols. Cancer Radiother. 2019 Dec;23(8):874-882. doi: 10.1016/j.canrad.2019.09.002. Epub 2019 Oct 11. PMID 31611051
- [Background] Strnad V, Major T, Polgar C, Lotter M, Guinot JL, Gutierrez-Miguelez C, Galalae R, Van Limbergen E, Guix B, Niehoff P, Lossl K, Hannoun-Levi JM. ESTRO-ACROP guideline: Interstitial multi-catheter breast brachytherapy as Accelerated Partial Breast Irradiation alone or as boost - GEC-ESTRO Breast Cancer Working Group practical recommendations. Radiother Oncol. 2018 Sep;128(3):411-420. doi: 10.1016/j.radonc.2018.04.009. Epub 2018 Apr 21. PMID 29691075
- [Background] Shah C, Vicini F, Shaitelman SF, Hepel J, Keisch M, Arthur D, Khan AJ, Kuske R, Patel R, Wazer DE. The American Brachytherapy Society consensus statement for accelerated partial-breast irradiation. Brachytherapy. 2018 Jan-Feb;17(1):154-170. doi: 10.1016/j.brachy.2017.09.004. Epub 2017 Oct 23. PMID 29074088
- [Background] Lancellotta V, Seipelt L, Hannoun-Levi JM, Tagliaferri L, Chand ME, Perrucci E, Valentini V, Aristei C, Kovacs G, Soror T. Multi-institutional evaluation of the reproducibility and the accuracy of the objective breast cosmesis scale. Brachytherapy. 2018 Nov-Dec;17(6):944-948. doi: 10.1016/j.brachy.2018.07.016. Epub 2018 Aug 24. PMID 30150016
- [Background] Correa C, Harris EE, Leonardi MC, Smith BD, Taghian AG, Thompson AM, White J, Harris JR. Accelerated Partial Breast Irradiation: Executive summary for the update of an ASTRO Evidence-Based Consensus Statement. Pract Radiat Oncol. 2017 Mar-Apr;7(2):73-79. doi: 10.1016/j.prro.2016.09.007. Epub 2016 Sep 17. PMID 27866865
- [Background] Polgar C, Ott OJ, Hildebrandt G, Kauer-Dorner D, Knauerhase H, Major T, Lyczek J, Guinot JL, Dunst J, Miguelez CG, Slampa P, Allgauer M, Lossl K, Polat B, Kovacs G, Fischedick AR, Fietkau R, Resch A, Kulik A, Arribas L, Niehoff P, Guedea F, Schlamann A, Potter R, Gall C, Uter W, Strnad V; Groupe Europeen de Curietherapie of European Society for Radiotherapy and Oncology (GEC-ESTRO). Late side-effects and cosmetic results of accelerated partial breast irradiation with interstitial brachytherapy versus whole-breast irradiation after breast-conserving surgery for low-risk invasive and in-situ carcinoma of the female breast: 5-year results of a randomised, controlled, phase 3 trial. Lancet Oncol. 2017 Feb;18(2):259-268. doi: 10.1016/S1470-2045(17)30011-6. Epub 2017 Jan 14. PMID 28094198
- [Background] Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. November 27, 2017. Access: https://ctep.cancer.gov/protocoldevelopment/electronic_applications/ctc.htm#ctc_50
- [Background] Vicini F, Shah C, Tendulkar R, Wobb J, Arthur D, Khan A, Wazer D, Keisch M. Accelerated partial breast irradiation: An update on published Level I evidence. Brachytherapy. 2016 Sep-Oct;15(5):607-15. doi: 10.1016/j.brachy.2016.06.007. Epub 2016 Jul 27. PMID 27475478
- [Background] Strnad V, Ott OJ, Hildebrandt G, Kauer-Dorner D, Knauerhase H, Major T, Lyczek J, Guinot JL, Dunst J, Gutierrez Miguelez C, Slampa P, Allgauer M, Lossl K, Polat B, Kovacs G, Fischedick AR, Wendt TG, Fietkau R, Hindemith M, Resch A, Kulik A, Arribas L, Niehoff P, Guedea F, Schlamann A, Potter R, Gall C, Malzer M, Uter W, Polgar C; Groupe Europeen de Curietherapie of European Society for Radiotherapy and Oncology (GEC-ESTRO). 5-year results of accelerated partial breast irradiation using sole interstitial multicatheter brachytherapy versus whole-breast irradiation with boost after breast-conserving surgery for low-risk invasive and in-situ carcinoma of the female breast: a randomised, phase 3, non-inferiority trial. Lancet. 2016 Jan 16;387(10015):229-38. doi: 10.1016/S0140-6736(15)00471-7. Epub 2015 Oct 19. PMID 26494415
- [Background] Brierley JD, Gospodarowicz MK, Wittekind C (Editors). (AJCC) TNM Classification of Malignant Tumours, 8th Edition. 2016, Wiley-Blackwell, www.wiley.com
- [Background] Strnad V, Hannoun-Levi JM, Guinot JL, Lossl K, Kauer-Dorner D, Resch A, Kovacs G, Major T, Van Limbergen E; Working Group Breast Cancer of GEC-ESTRO. Recommendations from GEC ESTRO Breast Cancer Working Group (I): Target definition and target delineation for accelerated or boost Partial Breast Irradiation using multicatheter interstitial brachytherapy after breast conserving closed cavity surgery. Radiother Oncol. 2015 Jun;115(3):342-8. doi: 10.1016/j.radonc.2015.06.010. Epub 2015 Jun 20. PMID 26104975
- [Background] Perrucci E, Lancellotta V, Bini V, Falcinelli L, Farneti A, Margaritelli M, Capezzali G, Palumbo I, Aristei C. Quality of life and cosmesis after breast cancer: whole breast radiotherapy vs partial breast high-dose-rate brachytherapy. Tumori. 2015 Mar-Apr;101(2):161-7. doi: 10.5301/tj.5000233. Epub 2015 Mar 11. PMID 25768319
- [Background] Cardoso MJ, Oliveira H, Cardoso J. Assessing cosmetic results after breast conserving surgery. J Surg Oncol. 2014 Jul;110(1):37-44. doi: 10.1002/jso.23596. Epub 2014 Mar 13. PMID 24623360
- [Background] Polgar C, Fodor J, Major T, Sulyok Z, Kasler M. Breast-conserving therapy with partial or whole breast irradiation: ten-year results of the Budapest randomized trial. Radiother Oncol. 2013 Aug;108(2):197-202. doi: 10.1016/j.radonc.2013.05.008. Epub 2013 Jun 3. PMID 23742961
- [Background] Cardoso MJ, Cardoso JS, Vrieling C, Macmillan D, Rainsbury D, Heil J, Hau E, Keshtgar M. Recommendations for the aesthetic evaluation of breast cancer conservative treatment. Breast Cancer Res Treat. 2012 Oct;135(3):629-37. doi: 10.1007/s10549-012-1978-8. Epub 2012 Feb 4. PMID 22307267
- [Background] Polgar C, Van Limbergen E, Potter R, Kovacs G, Polo A, Lyczek J, Hildebrandt G, Niehoff P, Guinot JL, Guedea F, Johansson B, Ott OJ, Major T, Strnad V; GEC-ESTRO breast cancer working group. Patient selection for accelerated partial-breast irradiation (APBI) after breast-conserving surgery: recommendations of the Groupe Europeen de Curietherapie-European Society for Therapeutic Radiology and Oncology (GEC-ESTRO) breast cancer working group based on clinical evidence (2009). Radiother Oncol. 2010 Mar;94(3):264-73. doi: 10.1016/j.radonc.2010.01.014. Epub 2010 Feb 22. PMID 20181402
- [Background] Stevens MJ, Cooper SG, Cross P, Wang Y. Accelerated partial breast irradiation using interstitial high dose rate iridium brachytherapy: Early Australian experience and review of the literature. Australas Radiol. 2006 Apr;50(2):143-51. doi: 10.1111/j.1440-1673.2006.01558.x. PMID 16635033
- [Background] Kuske RR, Winter K, Arthur DW, Bolton J, Rabinovitch R, White J, Hanson W, Wilenzick RM. Phase II trial of brachytherapy alone after lumpectomy for select breast cancer: toxicity analysis of RTOG 95-17. Int J Radiat Oncol Biol Phys. 2006 May 1;65(1):45-51. doi: 10.1016/j.ijrobp.2005.11.027. Epub 2006 Feb 28. PMID 16503383
- [Background] Wazer DE, Kaufman S, Cuttino L, DiPetrillo T, Arthur DW. Accelerated partial breast irradiation: an analysis of variables associated with late toxicity and long-term cosmetic outcome after high-dose-rate interstitial brachytherapy. Int J Radiat Oncol Biol Phys. 2006 Feb 1;64(2):489-95. doi: 10.1016/j.ijrobp.2005.06.028. Epub 2005 Oct 24. PMID 16246495
- [Background] Taghian AG, Recht A. Update on accelerated partial-breast irradiation. Curr Oncol Rep. 2006 Jan;8(1):35-41. doi: 10.1007/s11912-006-0007-7. PMID 16464401
- [Background] Chen PY, Vicini FA, Benitez P, Kestin LL, Wallace M, Mitchell C, Pettinga J, Martinez AA. Long-term cosmetic results and toxicity after accelerated partial-breast irradiation: a method of radiation delivery by interstitial brachytherapy for the treatment of early-stage breast carcinoma. Cancer. 2006 Mar 1;106(5):991-9. doi: 10.1002/cncr.21681. PMID 16421922
- [Background] Vicini FA, Arthur DW. Breast brachytherapy: North American experience. Semin Radiat Oncol. 2005 Apr;15(2):108-15. doi: 10.1016/j.semradonc.2004.10.005. PMID 15809936
- [Background] Arthur DW, Vicini FA. Accelerated partial breast irradiation as a part of breast conservation therapy. J Clin Oncol. 2005 Mar 10;23(8):1726-35. doi: 10.1200/JCO.2005.09.045. No abstract available. PMID 15755981
- [Background] Cuttino LW, Todor D, Arthur DW. CT-guided multi-catheter insertion technique for partial breast brachytherapy: reliable target coverage and dose homogeneity. Brachytherapy. 2005;4(1):10-7. doi: 10.1016/j.brachy.2004.11.002. PMID 15737901
- [Background] Ott OJ, Schulz-Wendtland R, Uter W, Pfahlberg A, Beckmann MW, Sauer R, Strnad V. Fat necrosis after conserving surgery and interstitial brachytherapy and/or external-beam irradiation in women with breast cancer. Strahlenther Onkol. 2005 Oct;181(10):638-44. doi: 10.1007/s00066-005-1439-y. PMID 16220402
- [Background] Major T, Fodor J, Takacsi-Nagy Z, Agoston P, Polgar C. Evaluation of HDR interstitial breast implants planned by conventional and optimized CT-based dosimetry systems with respect to dose homogeneity and conformality. Strahlenther Onkol. 2005 Feb;181(2):89-96. doi: 10.1007/s00066-005-1350-6. PMID 15702297
- [Background] Sarin R. Partial-breast treatment for early breast cancer: emergence of a new paradigm. Nat Clin Pract Oncol. 2005 Jan;2(1):40-7. doi: 10.1038/ncponc0071. PMID 16264855
- [Background] Vicini FA, Beitsch PD, Quiet CA, Keleher A, Garcia D, Snider HC, Gittleman MA, Zannis VJ, Kuerer H, Whitacre EB, Whitworth PW, Fine RE, Haffty BG, Arrambide LS. First analysis of patient demographics, technical reproducibility, cosmesis, and early toxicity: results of the American Society of Breast Surgeons MammoSite breast brachytherapy trial. Cancer. 2005 Sep 15;104(6):1138-48. doi: 10.1002/cncr.21289. PMID 16088962
- [Background] Weed DW, Edmundson GK, Vicini FA, Chen PY, Martinez AA. Accelerated partial breast irradiation: a dosimetric comparison of three different techniques. Brachytherapy. 2005;4(2):121-9. doi: 10.1016/j.brachy.2004.12.005. PMID 15893265
- [Background] Reitsamer R, Peintinger F, Sedlmayer F, Kopp M, Cimpoca W, Menzel C. Accelerated partial breast irradiation after conservative surgery for breast cancer. Ann Surg. 2005 Jul;242(1):147-8; author reply 148-9. doi: 10.1097/01.sla.0000169569.09715.c0. No abstract available. PMID 15973113
- [Background] Rivard MJ, Coursey BM, DeWerd LA, Hanson WF, Huq MS, Ibbott GS, Mitch MG, Nath R, Williamson JF. Update of AAPM Task Group No. 43 Report: A revised AAPM protocol for brachytherapy dose calculations. Med Phys. 2004 Mar;31(3):633-74. doi: 10.1118/1.1646040. PMID 15070264
- [Background] Strnad V, Ott O, Potter R, Hildebrandt G, Hammer J, Resch A, Lotter M, Ackermann S, Beckmann MW, Sauer R. Interstitial brachytherapy alone after breast conserving surgery: interim results of a German-Austrian multicenter phase II trial. Brachytherapy. 2004;3(3):115-9. doi: 10.1016/j.brachy.2004.08.003. PMID 15533801
- [Background] Rosenstein BS, Lymberis SC, Formenti SC. Biologic comparison of partial breast irradiation protocols. Int J Radiat Oncol Biol Phys. 2004 Dec 1;60(5):1393-404. doi: 10.1016/j.ijrobp.2004.05.072. PMID 15590170
- [Background] Makarewicz R (red.). Brachyterapia HDR. Via Medica. Gdańsk 2004.
- [Background] Das RK, Patel R, Shah H, Odau H, Kuske RR. 3D CT-based high-dose-rate breast brachytherapy implants: treatment planning and quality assurance. Int J Radiat Oncol Biol Phys. 2004 Jul 15;59(4):1224-8. doi: 10.1016/j.ijrobp.2004.03.030. PMID 15234059
- [Background] Kuerer HM, Julian TB, Strom EA, Lyerly HK, Giuliano AE, Mamounas EP, Vicini FA. Accelerated partial breast irradiation after conservative surgery for breast cancer. Ann Surg. 2004 Mar;239(3):338-51. doi: 10.1097/01.sla.0000114219.71899.13. PMID 15075650
- [Background] Van Limbergen E. Indications and technical aspects of brachytherapy in breast conserving treatment of breast cancer. Cancer Radiother. 2003 Apr;7(2):107-20. doi: 10.1016/s1278-3218(03)00015-5. PMID 12719040
- [Background] Arthur D. Accelerated partial breast irradiation: a change in treatment paradigm for early stage breast cancer. J Surg Oncol. 2003 Dec;84(4):185-91. doi: 10.1002/jso.10318. No abstract available. PMID 14756428
- [Background] Vicini FA et al. Limited-field radiation therapy in the management of early-stage breast cancer. J Natl Cancer Inst, 2003. 95(16): p. 1205-1210. Arthur DW, Koo D, Zwicker RD, et al. Partial Breast Brachytherapy Following Lumpectomy: a Low Dose Rate and High Dose Rate Experience. Int J Radiat Oncol Biol Phys 2003; 56:681-689.
- [Background] Arthur DW, Vicini FA, Kuske RR, Wazer DE, Nag S; American Brachytherapy Society. Accelerated partial breast irradiation: an updated report from the American Brachytherapy Society. Brachytherapy. 2003;2(2):124-30. doi: 10.1016/S1538-4721(03)00107-7. PMID 15062155
- [Background] Lawenda BD, Taghian AG, Kachnic LA, Hamdi H, Smith BL, Gadd MA, Mauceri T, Powell SN. Dose-volume analysis of radiotherapy for T1N0 invasive breast cancer treated by local excision and partial breast irradiation by low-dose-rate interstitial implant. Int J Radiat Oncol Biol Phys. 2003 Jul 1;56(3):671-80. doi: 10.1016/s0360-3016(03)00071-3. PMID 12788172
- [Background] Polgar C, Sulyok Z, Fodor J, Orosz Z, Major T, Takacsi-Nagy Z, Mangel LC, Somogyi A, Kasler M, Nemeth G. Sole brachytherapy of the tumor bed after conservative surgery for T1 breast cancer: five-year results of a phase I-II study and initial findings of a randomized phase III trial. J Surg Oncol. 2002 Jul;80(3):121-8; discussion 129. doi: 10.1002/jso.10110. PMID 12115793
- [Background] Wazer DE, Berle L, Graham R, Chung M, Rothschild J, Graves T, Cady B, Ulin K, Ruthazer R, DiPetrillo TA. Preliminary results of a phase I/II study of HDR brachytherapy alone for T1/T2 breast cancer. Int J Radiat Oncol Biol Phys. 2002 Jul 15;53(4):889-97. doi: 10.1016/s0360-3016(02)02824-9. PMID 12095554
- [Background] Vicini FA, Baglan KL, Kestin LL, Mitchell C, Chen PY, Frazier RC, Edmundson G, Goldstein NS, Benitez P, Huang RR, Martinez A. Accelerated treatment of breast cancer. J Clin Oncol. 2001 Apr 1;19(7):1993-2001. doi: 10.1200/JCO.2001.19.7.1993. PMID 11283132
- [Background] Wazer DE, Lowther D, Boyle T, Ulin K, Neuschatz A, Ruthazer R, DiPetrillo TA. Clinically evident fat necrosis in women treated with high-dose-rate brachytherapy alone for early-stage breast cancer. Int J Radiat Oncol Biol Phys. 2001 May 1;50(1):107-11. doi: 10.1016/s0360-3016(00)01541-8. PMID 11316552
- [Background] King TA, Bolton JS, Kuske RR, Fuhrman GM, Scroggins TG, Jiang XZ. Long-term results of wide-field brachytherapy as the sole method of radiation therapy after segmental mastectomy for T(is,1,2) breast cancer. Am J Surg. 2000 Oct;180(4):299-304. doi: 10.1016/s0002-9610(00)00454-2. PMID 11113440
- [Background] Nag S, Kuske RR, Vicini FA, Arthur DW, Zwicker RD. Brachytherapy in the treatment of breast cancer. Oncology (Williston Park). 2001 Feb;15(2):195-202, 205; discussion 205-7. doi: 10.1016/s0167-8140(01)80063-3. PMID 11252933
- [Background] Polgar C, Major T, Somogyi A, Fodor J, Toth J, Sulyok Z, Forrai G, Takacsi-Nagy Z, Mangel LC, Nemeth G. Sole brachytherapy of the tumor bed after breast conserving surgery: a new radiotherapeutic strategy for patients at low risk of local relapse. Neoplasma. 1999;46(3):182-9. PMID 10613595
- [Background] Vicini F, Kini VR, Chen P, Horwitz E, Gustafson G, Benitez P, Edmundson G, Goldstein N, McCarthy K, Martinez A. Irradiation of the tumor bed alone after lumpectomy in selected patients with early-stage breast cancer treated with breast conserving therapy. J Surg Oncol. 1999 Jan;70(1):33-40. doi: 10.1002/(sici)1096-9098(199901)70:13.0.co;2-o. PMID 9989418
- [Background] Kuske RR Jr. Breast brachytherapy. Hematol Oncol Clin North Am. 1999 Jun;13(3):543-58, vi-vii. doi: 10.1016/s0889-8588(05)70074-5. PMID 10432428
- [Background] Nath R, Anderson LL, Luxton G, Weaver KA, Williamson JF, Meigooni AS. Dosimetry of interstitial brachytherapy sources: recommendations of the AAPM Radiation Therapy Committee Task Group No. 43. American Association of Physicists in Medicine. Med Phys. 1995 Feb;22(2):209-34. doi: 10.1118/1.597458. No abstract available. PMID 7565352
- [Background] Cox JD, Stetz J, Pajak TF. Toxicity criteria of the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC). Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1341-6. doi: 10.1016/0360-3016(95)00060-C. No abstract available. PMID 7713792
- [Background] Harris JR, Levene MB, Svensson G, Hellman S. Analysis of cosmetic results following primary radiation therapy for stages I and II carcinoma of the breast. Int J Radiat Oncol Biol Phys. 1979 Feb;5(2):257-61. doi: 10.1016/0360-3016(79)90729-6. No abstract available. PMID 110740